CLINICAL TRIAL: NCT06876363
Title: A Phase 1/2 Open-Label, Single-Ascending-Dose Study of EN-374, a Helper-Dependent Adenoviral-Based Gene Therapy, in Participants With X-Linked Chronic Granulomatous Disease
Brief Title: Study of EN-374 Gene Therapy in Participants With X-Linked Chronic Granulomatous Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ensoma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN-374-101
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: X-Linked Chronic Granulomatous Disease
Keywords: CGD; X-CGD; Chronic Granulomatous Disease; X-Linked Chronic Granulomatous Disease; Granulomatous Disease, Chronic; Genetic Therapy; Gene Therapy; in vivo Gene Therapy; Gene Addition Therapy; in vivo Gene Addition Therapy; Hematopoietic Stem Cell Gene Therapy; in vivo Hematopoietic Stem Cell Gene Therapy
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EN-374 (Experimental): Single dose of EN-374 administered by intravenous infusion after mobilization and followed by enrichment
  Interventions: Genetic: EN-374

INTERVENTIONS:
Genetic: EN-374 — Single dose of EN-374 administered by intravenous infusion after mobilization and followed by enrichment

SUMMARY:
The goal of this clinical trial is to evaluate the safety and potential efficacy of the EN-374 treatment regimen and identify a dose level for further evaluation in participants with x-linked chronic granulomatous disease.

The main questions it aims to answer are:

* safety of the EN-374 treatment regimen
* effect of the EN-374 treatment regimen on the production of functional neutrophils with NADPH oxidase activity

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is a rare primary immune deficiency disorder characterized by recurrent bacterial or fungal infections starting in infancy. The x-linked form of CGD (X-CGD) is caused by mutations in the CYBB gene.

EN-374 is a helper-dependent adenoviral (HDAd)-based gene therapy in development for the treatment of X-CGD using an in vivo approach, which is administered by IV infusion, to genetically modify hematopoietic stem cells (HSCs) to express a wild-type CYBB gene. The EN-374 treatment regimen includes HSC mobilization, immune prophylaxis, EN-374 administration, and enrichment of genetically modified HSCs.

Adult participants with X-CGD will be enrolled into the dose-escalation part of the study. Following completion of the adult cohorts, then pediatric participants will be enrolled into the dose-expansion part of the study in decreasing age cohorts from ≥ 12 and < 18 years of age, to ≥ 2 and < 12 years of age, and finally to ≥ 3 months and < 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥ 18 years of age during dose escalation, then ≥ 3 months of age during dose expansion
* Diagnosis of X-CGD with DHR+ cells ≤ 5% and a pathogenic mutation in the CYBB gene
* History of at least 1 severe infection requiring medical intervention or chronic inflammatory disorder
* Does not have a suitable, available, and willing human leukocyte antigens (HLA)-matched (10/10) related donor
* Non-sterile male participants who are or may become sexually active with female partners of childbearing potential are required to use highly effective contraception
* Informed consent, with informed assent from capable participants
* Adequate organ function

Exclusion Criteria:

* Active bacteremia or fungemia
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* History or clinical evidence of any medical or social issues likely to put the participant at additional risk or to interfere with study conduct
* History of HSCT or granulocyte transfusions
* Known hypersensitivity to elements in the treatment regimen
* Undergone investigational gene therapy
* Treated with another investigational drug product within 30 days before screening
* Unable to comply with the visits and requirements of the protocol as determined by the Investigator

Min Age: 3 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety of EN-374 | From start of mobilization until Month 12
  Incidence rate across all age groups of:
  * treatment-emergent adverse events (TEAEs)
  * treatment-related TEAEs (TRAEs)
  * serious adverse events (SAEs)

SECONDARY OUTCOMES:
Effect of the EN-374 treatment regimen on the production of functional neutrophils with NADPH oxidase activity | From infusion of EN-374 until Month 12
  * Change from baseline in the percentage of dihydrorhodamine (DHR)+ neutrophils
  * Change from baseline in the percentage of participants with ≥ 10%, 20%, 30%, 40%, or 50% DHR+ neutrophils

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Irving Medical Center, Morgan Stanley Children's Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - University of Utah, Primary Children's Hospital, Salt Lake City, Utah